CLINICAL TRIAL: NCT03531619
Title: Dizziness and Neck Pain - is There a Relationship and Does it Matter?
Brief Title: The Relationship Between Dizziness and Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/783
Record Dates: First submitted 2018-03-12; First posted 2018-05-22 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Dizziness; Vertigo; Neck Pain
Keywords: posturography; quality of life; pressure algometry; cervicogenic dizziness
MeSH Terms: conditions — Dizziness; Vertigo; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Dizziness: Patients referred to a neuro-otological clinic due to dizziness who answer that they do not suffer from neck pain
- Dizziness and neck pain: Patients referred to a neuro-otological clinic due to dizziness who answer that they suffer from neck pain
- Neck pain: Patients referred to a rehabilitation center due to neck pain who answer that they do not suffer from dizziness
- Neck pain and dizziness: Patients referred to a rehabilitation center due to neck pain who answer that the suffer from dizziness
- Healthy Control: Healthy Controls without neck pain or dizziness

SUMMARY:
Both dizziness and neck pain are common complaints in the Norwegian population. The cervical spine has a highly developed proprioceptive system, which is involved in head and gaze stabilization as well as postural control. Thus, it has been argued that dizziness and/or unsteadiness can occur due to loss of or inadequate stimulation of neck receptors in patients with neck pain. Still, the notion of dizziness due to cervical dysfunction is a controversial topic. However, clinicians report that patients referred for dizziness often complain of neck pain, and vice versa.

This study is a multi-center study including patients referred to 1) a neuro-otologic clinic due to dizziness and 2) a rehabilitation clinic due to neck pain. Both clinics are tertiary care university clinics. The study explores the prevalence, severity and spectrum of symptoms as well as clinical findings in patients with various combinations of dizziness and neck pain. The aim is to see if these patient groups differ from each other in terms of clinical characteristics, symptoms and quality of life. Additionally, the aim is to examine if there is a relationship between neck dysfunction and dizziness, and last, if the symptoms persist longer in patients with both dizziness and neck pain.

DETAILED DESCRIPTION:
This is a longitudinal study with data collected at baseline, 6 months and 3 years follow-up.

Variables collected at baseline include age, sex, symptom variables including Dizziness Handicap Inventory, Vertigo Symptom Scale Short Form, Haukeland Dizziness Questionnaire, Visual analog scale, Hospital Anxiety and Depression Scale, RAND-12, dynamic posturography, video-based head impulse test, bithermal caloric tests, Neck Disability Index, as well as neck examinations including pressure algometry and measurements of the range of neck movements.

Follow-up data after 6 months include the same patient-reported outcomes as at baseline.

ELIGIBILITY:
Inclusion criteria for patients:

* Residence within the Health Region of Western Norway AND
* Referral to the ENT department of Haukeland University Hospital due to vertigo OR
* Referral to Nordås Outpatient Clinic due to neck pain lasting > 3 months

Exclusion criteria for patients:

* Severe orthopaedic or neurologic disease affecting postural balance
* Inability to undergo test protocol due to physical or language barriers
* Quaternary referrals (vestibular schwannomas or divers with vestibular disorders)

Inclusion criteria for healthy controls:

- Employees at Haukeland University Hospital

Exclusion criteria for healthy controls:

* Known neurologic or vestibular disease or ongoing ear disease.
* Neck pain within last 3 months

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients referred to the ENT department of Haukeland University Hospital due to vertigo with suspected vestibular origin will be divided into two groups depending on whether or not they report concurrent neck pain.
  2. Patients referred to the Nordås clinic due to chronic neck pain will be divided into two groups depending on whether or not the report concurrent dizziness.
  The healthy controls will be recruited among employees at Haukeland University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference between Groups in the Dizziness Handicap Inventory (DHI) | Baseline and 6 months follow-up
  25-item symptom score. 0-100 Points on dizziness handicap severity
Difference betwee Groups in the Neck Disability Index (NDI) | Baseline and 6 months follow-up
  10-time symptom score. 0-50 Points on neck disabilty severity

SECONDARY OUTCOMES:
Correlation between Posturography and neck pain | Baseline
  Path length is used as measure of steadiness. Neck pain is measured With a pressure algometer, measuring the pressure pain threshold of the neck in kilo pascal.

CONTACTS AND LOCATIONS:
Overall Officials: Stein Helge Glad Nordhal, Professor II, Study Director — Norwegian National Advisory Unit on Vestibular Disorders
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Knapstad MK, Goplen FK, Ask T, Skouen JS, Nordahl SHG. Associations between pressure pain threshold in the neck and postural control in patients with dizziness or neck pain - a cross-sectional study. BMC Musculoskelet Disord. 2019 Nov 10;20(1):528. doi: 10.1186/s12891-019-2922-4. PMID 31707980